CLINICAL TRIAL: NCT01777555
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled Study Investigating the Efficacy and Safety of Inhaled CVT 301 (Levodopa Inhalation Powder) in Parkinson's Disease Patients With Motor Response Fluctuations (OFF Phenomena)
Brief Title: Efficacy and Safety Study of Inhaled CVT 301 in Parkinson's Disease Patients for Treatment of OFF Episodes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVT-301-003; 2012-005822-31 (EudraCT Number)
Record Dates: First submitted 2013-01-23; First posted 2013-01-29 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2015-05

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Parkinson's Disease; Motor fluctuations; levodopa; inhaled drugs; Off episodes
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CVT-301 (Experimental): CVT-301 at Dose Level 1 for 1st 14 days of treatment then increased to Dose level 2 for last 14 days of treatment.
  Interventions: Drug: CVT-301
- Inhaled Placebo (Placebo Comparator): Subjects randomized to receive placebo in a 1:1 randomization scheme
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CVT-301
  Other Names: Levodopa Inhalation Powder
  Arms: CVT-301
Drug: Placebo
  Arms: Inhaled Placebo

SUMMARY:
This randomized, multicenter, placebo-controlled, double-blind study will evaluate the efficacy and safety of inhaled CVT 301 compared with placebo in PD patients experiencing motor response fluctuations (OFF phenomena) as an outpatient (i.e., at home) and in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's Disease (PD) diagnosed between the ages of 30 and 80 years;
* Hoehn and Yahr Stage 1-3 in an "on" state;
* Require levodopa-containing medication regimen at least 4 times during the waking day;
* Experience motor fluctuations with a minimum of 2 hours of average daily "off" time per waking day (excluding early morning "off" time) and demonstrate levodopa responsiveness;
* Are on stable PD medication regimen.

Exclusion Criteria:

* Pregnant or lactating females;
* Previous surgery for PD or plan to have stereotactic surgery during the study period;
* History of psychotic symptoms requiring treatment, or suicide ideation or attempt within last year;
* Adequate lung function as measured by spirometry;
* Any significant condition, severe concurrent disease, abnormality or finding that would make patients unsuitable or may compromise patient safety.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in average Unified Parkinson's Disease Rating Scale Part III motor score | pre-dose to 60 minutes following treatment

SECONDARY OUTCOMES:
Time to resolution of OFF episode to an ON state. | 28 days duration outpatient treatment
To characterize the safety (including pulmonary safety)of CVT-301 when used chronically to provide relief from OFF episodes. | change from baseline through 28 days outpatient use
  Adverse experiences, ECGs, vital signs, clinical laboratory evaluation, pulmonary function using spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Martin Freed, MD, Study Chair — Acorda Therapeutics
Locations (22):
- United States (13):
  - Civitas Investigational Site 1013, Little Rock, Arkansas
  - Civitas Investigational Site 1004, Boca Raton, Florida
  - Civitas Investigational Site 1002, Port Charlotte, Florida
  - Civitas Investigational Site 1015, Tampa, Florida
  - Civitas Investigational Site 1007, Kansas City, Kansas
  - Civitas Investigational Site 1010, Boston, Massachusetts
  - Civitas Investigational Site 1001, Bingham Farms, Michigan
  - Civitas Investigational Site 1008, Roseville, Michigan
  - Civitas Investigational Site 1009, Saint Louis, Michigan
  - Civitas Investigational Site 1005, West Bloomfield, Michigan
  - Civitas Investigational Site 1011, Kingston, New York
  - Civitas Investigational Site 1014, Cleveland, Ohio
  - Civitas Investigational Site 1003, Kirkland, Washington
- Italy (3):
  - Civitas Investigational Site 4003, Cassino
  - Civitas Investigational Site 4002, Chieti
  - Civitas Investigational Site 4001, Rome
- Serbia (2):
  - Civitas Investigational Site 3001, Belgrade
  - Civitas Investigational Site 3002, Belgrade
- United Kingdom (4):
  - Civitas Investigational Site 2004, Cambridge
  - Civitas Investigational Site 200, Glasgow
  - Civitas Investigational Site 2001, London
  - Civitas Investigational Site 2003, Stoke-on-Trent